CLINICAL TRIAL: NCT03708198
Title: Pharmacokinetics of Single-Dose Liposomal Bupivacaine in Surgeon Performed Intercostal Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, William Manson, MD, Assistant Professor of Anesthesiology, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 180006
Record Dates: First submitted 2018-06-08; First posted 2018-10-17 (Actual); Results first posted 2022-05-23 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Thoracic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intercostal Nerve Block (Other): The study participants will be given a standard 266 mg single dose injection of liposomal bupivacaine by the surgeon at the start of the surgery.
  Interventions: Drug: Liposomal Bupivacaine

INTERVENTIONS:
Drug: Liposomal Bupivacaine — intercostal block

SUMMARY:
Post-surgery pain management is critical for ensuring timely patient recovery and minimizing complications. Part of the multimodal approach to managing severe acute pain in the days following surgeries is the use of nerve blocks. The relatively short-lived effect of commonly used local anesthetics recently prompted the development and subsequent approval of a liposomal formulation of bupivacaine (Exparel; Pacira Pharmaceuticals, Parsippany, New Jersey). It has demonstrated favorable pharmacokinetics compared to bupivacaine HCl(hydrochloride), with a slower release into blood stream of up to 96 hours after administration, following a single dose wound infiltration at the end of various surgeries. Studies using other modes of administration reported similar results.

Thoracic surgeries pose an exceptional challenge as they are one of the most painful surgeries and poor pain-management contributes to reduced quality of life and severely delayed recovery. The anesthesiology protocol within the Enhanced Recovery After Surgery (ERAS) program at medical centers across the world aim to increase patient comfort after surgery while reducing complications and use of opioids. As a common part of this protocol, intercostal nerve blocks with liposomal bupivacaine are regularly utilized for reduction of post-thoracotomy pain and studies show that it may be just as or more effective than bupivacaine HCl for treatment of pain, decreasing hospital stays and reducing the incidence of complications.

Despite its frequent use in the surgical room for nerve blocks, the pharmacokinetics of a single dose injection of liposomal bupivacaine at the intercostal nerves has never been investigated. The aim of this study is to assess the pharmacokinetics of liposomal bupivacaine injected at the intercostal nerves. The results of this small-scale study will aid in the development of larger such studies in the future, and may aid in the standardization of post-thoracotomy pain management. Specifically, the information gleaned from this study will allow for the optimal use of additional local anesthetics, particularly those administered intravenously, for the purpose of obtaining maximal pain relief while minimizing the occurrence of local anesthetic toxicity.

DETAILED DESCRIPTION:
In this study, patients who are undergoing thoracotomies will be consented separately from the surgery itself.

Patients will be consented for the study in the surgical clinic or on the day of the surgery in the Surgical Admission Suites (SAS), prior to being taken to the OR. The study participants will be given a standard 266 mg single dose injection of liposomal bupivacaine by the surgeon at the start of the surgery. Immediately prior to the injection of the local anesthetic, 5 ml of blood will be drawn from the patient via the arterial line. The arterial line will be placed as part of standard surgery procedure and not for the purposes of the study. Blood will then be drawn from the patient after the injection of the local anesthetic at 5 mins, 15 mins, 30 mins, 1, 2, 4, 8, 12, 24, 48, 72 and 96 h. Each blood draw will be 5 ml. Blood will be drawn a total of 13 times.

The arterial line will not remain in the patient for the purposes of the study and will be removed per standard procedure. If more blood samples are needed after the arterial line is removed, we will first attempt to obtain blood an existing venous catheter. If blood cannot be obtained this way, a venipuncture will be performed.

Blood samples will be analyzed for the following pharmacokinetic parameters: area under the serum concentration-time infinity (AUC), maximum observed serum concentration (Cmax), time to attain Cmax (Tmax), and apparent terminal elimination half-life (T1/2).

At the time blood samples are drawn, pain scores will be recorded on a standard ten-point pain scale. These pain scores will be omitted if the patient is under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* Undergoing thoracotomy

Exclusion Criteria:

* Non-English speaking
* Pregnant women (self reported)
* Prisoners
* Weighing <50 kg
* Allergy to local anesthetics
* Unable to consent for themselves

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2020-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Manson, MD, Principal Investigator — UVA Department of Anesthesiology
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu D, Onel E, Singla N, Kramer WG, Hadzic A. Pharmacokinetic profile of liposome bupivacaine injection following a single administration at the surgical site. Clin Drug Investig. 2013 Feb;33(2):109-15. doi: 10.1007/s40261-012-0043-z. PMID 23229686
- [Background] Davidson EM, Barenholz Y, Cohen R, Haroutiunian S, Kagan L, Ginosar Y. High-dose bupivacaine remotely loaded into multivesicular liposomes demonstrates slow drug release without systemic toxic plasma concentrations after subcutaneous administration in humans. Anesth Analg. 2010 Apr 1;110(4):1018-23. doi: 10.1213/ANE.0b013e3181d26d2a. PMID 20357145
- [Background] De Cosmo G, Aceto P, Gualtieri E, Congedo E. Analgesia in thoracic surgery: review. Minerva Anestesiol. 2009 Jun;75(6):393-400. Epub 2008 Oct 27. PMID 18953284
- [Background] Mehran RJ, Walsh GL, Zalpour A, Cata JP, Correa AM, Antonoff MB, Rice DC. Intercostal Nerve Blocks With Liposomal Bupivacaine: Demonstration of Safety, and Potential Benefits. Semin Thorac Cardiovasc Surg. 2017 Winter;29(4):531-537. doi: 10.1053/j.semtcvs.2017.06.004. Epub 2017 Jun 6. PMID 29698654
- [Background] Rice DC, Cata JP, Mena GE, Rodriguez-Restrepo A, Correa AM, Mehran RJ. Posterior Intercostal Nerve Block With Liposomal Bupivacaine: An Alternative to Thoracic Epidural Analgesia. Ann Thorac Surg. 2015 Jun;99(6):1953-60. doi: 10.1016/j.athoracsur.2015.02.074. Epub 2015 Apr 23. PMID 25912739

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intercostal Nerve Block
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intercostal Nerve Block
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 67 [21 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 15
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Tmax, or the Time Until the Maximum Concentration
Description: the tmax, or the time until the maximum concentration
Time Frame: until study completion, which is 6 months on average
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Intercostal Nerve Block
Number analyzed (Participants) | 15
Hours | 24 [12 to 36]

ADVERSE EVENTS:
Time Frame: six months
Description: The definition of adverse events or serious adverse events does not differ from the clinicaltrials.gov definition.
Arm/Group | Intercostal Nerve Block
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/98/NCT03708198/Prot_SAP_000.pdf